CLINICAL TRIAL: NCT00708227
Title: Pharmacogenetics of b2-Agonists in Asthma.
Status: Completed | Type: Observational
Sponsor: Nemours Children's Clinic (Other)
Collaborators: University of Florida (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kathryn Blake, PharmD, Senior Research Scientist, Nemours Children's Clinic
Other Study IDs: 82211; K23HL081245 (NIH)
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Results first posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Asthma
Keywords: Asthma; Pharmacogenetics; Salmeterol; African American; White
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The purpose of the epigenetic substudy is to collecting blood is for exploratory research into epigenetic effects of salmeterol therapy. Blood was collected at Visit 2 and Visit 3.
  Steps:
  * Obtain informed consent
  * Label vacutainer tube with patient's study ID number, visit number, date of collection (use a sharpee pen)
  * Collect 10mL blood sample into purple top tube before starting methacholine challenge (must be done before any albuterol is given at the visit)
  * Immediately place tube in crushed ice or in refrigerator
  * Spin tube; freeze tube with cells for future genotyping/methylation studies; divide plasma as equally as possible between the 3 cryotubes, freeze the EDTA tube and 3 cryotubes.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Whites ADRB2:ARG16ARG: All participants receive fluticasone for 2-weeks followed by fluticasone / salmeterol for 2-weeks at a dose commensurate with baseline inhaled corticosteroid dose. All participants receive ipratropium bromide for symptom rescue therapy.
- Whites ADRB2:GLY16GLY: All participants receive fluticasone for 2-weeks followed by fluticasone / salmeterol for 2-weeks at a dose commensurate with baseline inhaled corticosteroid dose. All participants receive ipratropium bromide for symptom rescue therapy.
- African American ADRB2:ARG16ARG: All participants receive fluticasone for 2-weeks followed by fluticasone / salmeterol for 2-weeks at a dose commensurate with baseline inhaled corticosteroid dose. All participants receive ipratropium bromide for symptom rescue therapy.
- African American ADRB2:GLY16GLY: All participants receive fluticasone for 2-weeks followed by fluticasone / salmeterol for 2-weeks at a dose commensurate with baseline inhaled corticosteroid dose. All participants receive ipratropium bromide for symptom rescue therapy.

SUMMARY:
This study will help to find out if having a certain genetic makeup influences how a person with asthma responds to salmeterol, one of the two drugs in Advair(R).

DETAILED DESCRIPTION:
Patients are being asked to take part in this research study because they have asthma. This clinical research study is being done to see if an asthmatic's gene make-up (DNA is made up of genes) affects the way they respond to a particular asthma medication called salmeterol. Certain genes make people tall or short. Certain genes give people brown or black hair. Similarly, certain genes may be associated with the way patients respond to asthma medications.

Salmeterol xinafoate (a long acting bronchodilator) and fluticasone propionate (an inhaled corticosteroid) are the medicines contained in Advair Diskus. During this study, patients with asthma will receive fluticasone inhaler (called Flovent) and Advair Diskus. The investigators want to find out if patients with asthma with certain genes respond in different ways to the salmeterol in Advair Diskus. The investigators also want to find out if patients with asthma with certain genes who are treated with salmeterol for two weeks have their airways open up less than usual when they use albuterol.

ELIGIBILITY:
Inclusion Criteria:

* Diplotype: Whites with specific diplotype and African Americans with specific diplotypes.
* Gender: Male or female. Women are eligible if they are not pregnant or lactating. Females subjects of childbearing potential will undergo a urine pregnancy test prior to each methacholine challenge test.
* Age: 10 years and older.
* Asthma Diagnosis: Physician diagnosed asthma according to American Thoracic Society criteria for at least 3 months.
* Asthma Therapy: There is no requirement for previous asthma therapy to be included in this study.
* Asthma Severity: forced expiratory volume in the first second (FEV1) must be >= 60% of predicted normal values for age, height, and gender.
* methacholine challenge test provocative concentration (20% fall in FEV1) of <=12]mg/ml.

Exclusion Criteria:

* History of life-threatening asthma: Any episode of asthma requiring intubation associated with hypercapnia, respiratory arrest, or hypoxic seizures.
* Asthma instability: Hospitalization for asthma within 3 months of Visit 1.
* Concurrent respiratory disease: Any respiratory disease other than asthma.
* Sensitivities: Sensitivities to methacholine, Flovent® MDI, ipratropium bromide, albuterol, or Advair Diskus® that would put the safety of the subject at risk.
* Respiratory Tract Infection: Any sinus, middle ear, oropharyngeal, upper or lower respiratory tract infection that has not resolved at least 2 weeks immediately preceding Visit 1, or for which antibiotic therapy has not been completed at least 2 weeks prior to Visit 1.
* Expected exposure to pollen allergen to which the patient is sensitive (by medical history of symptoms) during the 29 day study period. These patients can be studied when pollen exposure to which they are sensitive will not occur.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population was Whites and African Americans with specific ADRB2 diplotypes aged 10 years or older with physician diagnosed asthma according to American Thoracic Society criteria for at least 3 months, forced expiratory volume in the first second (FEV1) >= 60% of predicted normal values for age, height, and gender, and a methacholine challenge test provocative concentration (20% fall in FEV1) of <=12]mg/ml.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2007-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Blake, Pharm.D., Principal Investigator — Nemours Children's Clinic
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States

REFERENCES:
- [Result] Blake K, Cury JD, Hossain J, Tantisira K, Wang J, Mougey E, Lima J. Methacholine PC20 in African Americans and whites with asthma with homozygous genotypes at ADRB2 codon 16. Pulm Pharmacol Ther. 2013 Jun;26(3):342-7. doi: 10.1016/j.pupt.2013.01.009. Epub 2013 Feb 4. PMID 23384627

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Nemours Children's Health System, the University of Florida Jacksonville, health fairs and events, Edward Waters College, and from previous study participation. Participants were recruited between January 2008 and October 2011
Pre-assignment Details: Enrolled participants were excluded from receiving planned study treatment if they did not meet the ADRB2 genotype criteria and if they did not have a methacholine PC20 of 12.5mg/ml or less.
Groups:
- Whites ADRB2:ARG16ARG: All participants receive fluticasone for 2-weeks followed by fluticasone / salmeterol for 2-weeks at a dose commensurate with baseline inhaled corticosteroid dose. All participants receive ipratropium bromide for symptom rescue therapy.
  fluticasone: Fluticasone propionate MDI(dose to be determined by patient's current treatment) for 2 weeks, followed by Advair(R)Diskus (same dose of fluticasone propionate) for 2 weeks; Ipratropium bromide MDI used for prn symptom relief
- Whites ADRb2:GLY16GLY; African Americans ADRB2:ARG16ARG; African Americans ADRB2:GLY16GlY: All participants receive fluticasone for 2-weeks followed by fluticasone / salmeterol for 2-weeks at a dose commensurate with baseline inhaled corticosteroid dose. All participants receive ipratropium bromide for symptom rescue therapy.
  Salmeterol: Fluticasone propionate MDI(dose to be determined by patient's current treatment) for 2 weeks, followed by Advair(R)Diskus (same dose of fluticasone propionate) for 2 weeks; Ipratropium bromide MDI used for prn symptom relief
Period: Overall Study
Arm/Group | Whites ADRB2:ARG16ARG | Whites ADRb2:GLY16GLY | African Americans ADRB2:ARG16ARG | African Americans ADRB2:GLY16GlY
Started | 19 | 26 | 18 | 25
Completed | 18 | 21 | 17 | 22
Not Completed | 1 | 5 | 1 | 3
Not completed — Physician Decision | 0 | 3 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Whites ADRB2:ARG16ARG; African Americans ADRB2:ARG16ARG; African Americans ADRB2:GLY16GLY: All participants receive fluticasone for 2-weeks followed by fluticasone / salmeterol or 2-weeks at a dose commensurate with baseline inhaled corticosteroid dose. All participants receive ipratropium bromide for symptom rescue therapy.
  fluticasone: Fluticasone propionate MDI(dose to be determined by patient's current treatment) for 2 weeks, followed by Advair(R)Diskus (same dose of fluticasone propionate) for 2 weeks; Ipratropium bromide MDI used for prn symptom relief
- Whites ADRB2:GLY16GLY: All participants receive fluticasone for 2-weeks followed by fluticasone / salmeterol or 2-weeks at a dose commensurate with baseline inhaled corticosteroid dose. All participants receive ipratropium bromide for symptom rescue therapy.
  Salmeterol: Fluticasone propionate MDI(dose to be determined by patient's current treatment) for 2 weeks, followed by Advair(R)Diskus (same dose of fluticasone propionate) for 2 weeks; Ipratropium bromide MDI used for prn symptom relief
- Total: Total of all reporting groups
Arm/Group | Whites ADRB2:ARG16ARG | Whites ADRB2:GLY16GLY | African Americans ADRB2:ARG16ARG | African Americans ADRB2:GLY16GLY | Total
Number analyzed (Participants) | 19 | 26 | 18 | 25 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 6 | 9 | 10 | 30
  Between 18 and 65 years | 13 | 17 | 7 | 15 | 52
  >=65 years | 1 | 3 | 2 | 0 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (19) | 37 (20) | 27 (21) | 28 (17) | 32 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 13 | 18 | 61
  Male | 5 | 10 | 5 | 7 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 18 | 25 | 43
  White | 19 | 26 | 0 | 0 | 45
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 26 | 18 | 25 | 88
ADRB2 Genotype at Codon 16 [Count of Participants; unit: Participants] | 19 | 26 | 18 | 25 | 88

OUTCOME MEASURES:

1. Primary Outcome: Log10 PC20 to Methacholine After Visit 2
Description: Visit 2 log10 PC20 after receiving 2 weeks of Flovent
Time Frame: Visit 2:12 hours after last dose of Flovent
Population: All participants who had a methacholine challenge at Visit 2. All participants had received Flovent for 2 weeks.
Measure: Mean (Standard Deviation); unit: log10 mg/mL
Groups:
- Whites ADRB2:ARG16ARG: Log10 methacholine PC20 data in Whites with the ADRB2 ARG16ARG genotype after receiving 2 weeks of Flovent.
- Whites ADRB2:Gly16Gly: Log10 methacholine PC20 data in Whites with the ADRB2 GLY16GLY genotype after receiving 2 weeks of Flovent.
- African Americans ADRB2:ARG16ARG: Log10 methacholine PC20 data in African Americans with the ADRB2 ARG16ARG genotype after receiving 2 weeks of Flovent.
- African Americans ADRB2:GLY16GLY: Log10 methacholine PC20 data in African Americans with the ADRB2 GLY16GLY genotype after receiving 2 weeks of Flovent.
Arm/Group | Whites ADRB2:ARG16ARG | Whites ADRB2:Gly16Gly | African Americans ADRB2:ARG16ARG | African Americans ADRB2:GLY16GLY
Number analyzed (Participants) | 18 | 25 | 17 | 23
log10 mg/mL | 0.54 (0.65) | 0.48 (0.71) | 0.16 (0.57) | 0.53 (0.67)
Statistical Analysis 1: Comparison: Whites ADRB2:ARG16ARG vs Whites ADRB2:Gly16Gly vs African Americans ADRB2:ARG16ARG vs African Americans ADRB2:GLY16GLY; Test type: Superiority; p = 0.27, ANOVA

2. Primary Outcome: Log10 PC20 to Methacholine After Visit 3
Description: Visit 3 Log10 PC20 after receiving 2 weeks of Advair
Time Frame: Visit 3:12 hours after the last dose of Advair
Population: All participants who had a methacholine challenge at Visit 3. All participants had received Advair for 2 weeks.
Measure: Mean (Standard Deviation); unit: log10 mg/mL
Groups:
- Whites ADRB2:ARG16ARG: Visit 3 log10 methacholine PC20 data in Whites with the ADRB2 ARG16ARG genotype after receiving 2 weeks of Advair.
- Whites ADRB2:Gly16Gly: Visit 3 log10 methacholine PC20 data in Whites with the ADRB2 GLY16GLY genotype after receiving 2 weeks of Advair.
- African Americans ADRB2:ARG16ARG: Visit 3 log10 methacholine PC20 data in African Americans with the ADRB2 ARG16ARG genotype after receiving 2 weeks of Advair.
- African Americans ADRB2:GLY16GLY: Visit 3 log10 methacholine PC20 data in African Americans with the ADRB2 GLY16GLY genotype after receiving 2 weeks of Advair.
Arm/Group | Whites ADRB2:ARG16ARG | Whites ADRB2:Gly16Gly | African Americans ADRB2:ARG16ARG | African Americans ADRB2:GLY16GLY
Number analyzed (Participants) | 18 | 23 | 17 | 22
log10 mg/mL | 0.75 (0.65) | 0.78 (0.60) | 0.35 (0.63) | 0.75 (0.65)
Statistical Analysis 1: Comparison: Whites ADRB2:ARG16ARG vs Whites ADRB2:Gly16Gly vs African Americans ADRB2:ARG16ARG vs African Americans ADRB2:GLY16GLY; Test type: Superiority; p = 0.15, ANOVA

3. Primary Outcome: Log10 PC20 to Methacholine After Visit 4
Description: Visit 4 log10 PC20 to Methacholine after stopping Advair
Time Frame: 36 hours after the last dose of Advair
Population: All participants who had a methacholine challenge at Visit 4. All participants had discontinued Advair for 36 hours.
Measure: Mean (Standard Deviation); unit: log10 mg/mL
Groups:
- Whites ADRB2:ARG16ARG: Visit 4 log10 methacholine PC20 data in Whites with the ADRB2 ARG16ARG genotype after receiving 2 weeks of Flovent.
- Whites ADRB2:Gly16Gly: Visit 4 log10 methacholine PC20 data in Whites with the ADRB2 GLY16GLY genotype after receiving 2 weeks of Flovent.
- African Americans ADRB2:ARG16ARG: Visit 4 log10 methacholine PC20 data in African Americans with the ADRB2 ARG16ARG genotype after receiving 2 weeks of Flovent.
- African Americans ADRB2:GLY16GLY: Visit 4 log10 methacholine PC20 data in African Americans with the ADRB2 GLY16GLY genotype after receiving 2 weeks of Flovent.
Arm/Group | Whites ADRB2:ARG16ARG | Whites ADRB2:Gly16Gly | African Americans ADRB2:ARG16ARG | African Americans ADRB2:GLY16GLY
Number analyzed (Participants) | 18 | 21 | 17 | 22
log10 mg/mL | 0.73 (0.61) | 0.89 (0.57) | 0.36 (0.52) | 0.70 (0.66)
Statistical Analysis 1: Comparison: Whites ADRB2:ARG16ARG vs Whites ADRB2:Gly16Gly vs African Americans ADRB2:ARG16ARG vs African Americans ADRB2:GLY16GLY; Test type: Superiority; p = 0.06, ANOVA

4. Secondary Outcome: Bronchodilator Response to Methacholine (PC20) After Visit 2
Description: The area under the curve (AUC) bronchodilator response after Visit 2 methacholine challenge. 2.5mg of albuterol was administered at the time of maximal brochoconstriction once the methacholine PC20 was reached and the change in FEV1 was measured over the next 60 minutes post albuterol administration (bronchodilator response). FEV1 was measured at the following times: 0 (immediately upon completion of nebulization) and at 1, 3, 5, 10, 15, 20, 30, 45, and 60 minutes. Participants had received Flovent for 2 weeks at Visit 2.
Time Frame: 0 (immediately upon completion of nebulization) and at 1, 3, 5, 10, 15, 20, 30, 45, and 60 minutes after nebulization was complete which occurred 12 hours after the last dose of Flovent.
Population: All participants who had received Flovent for 2 weeks at Visit 2.
Measure: Mean (Standard Deviation); unit: Liters*min
Groups:
- Whites ADRB2:ARG16ARG; Whites ADRB2:Gly16Gly; African Americans ADRB2:ARG16ARG; African Americans ADRB2:GLY16GLY: The area under the curve (AUC) bronchodilator response after Visit 2 methacholine challenge. 2.5mg of albuterol was administered at the time of maximal brochoconstriction once the methacholine PC20 was reached. Participants had received Flovent for 2 weeks at Visit 2.
Arm/Group | Whites ADRB2:ARG16ARG | Whites ADRB2:Gly16Gly | African Americans ADRB2:ARG16ARG | African Americans ADRB2:GLY16GLY
Number analyzed (Participants) | 18 | 25 | 18 | 25
Liters*min | 188.5 (67.55) | 196.6 (63.3) | 169.9 (58.97) | 161.4 (42.7)

5. Secondary Outcome: Bronchodilator Response Following Methacholine Challenge at Visit 3
Description: The area under the curve (AUC) bronchodilator response after Visit 3 methacholine challenge. 2.5mg of albuterol was administered at the time of maximal brochoconstriction once the methacholine PC20 was reached and the change in FEV1 was measured over the next 60 minutes post albuterol administration (bronchodilator response). FEV1 was measured at the following times: 0 (immediately upon completion of nebulization) and at 1, 3, 5, 10, 15, 20, 30, 45, and 60 minutes. Participants had received Advair for 2 weeks at Visit 3.
Time Frame: 0 (immediately upon completion of nebulization) and at 1, 3, 5, 10, 15, 20, 30, 45, and 60 minutes after nebulization was complete which occurred 12 hours after the last dose of Advair
Population: The area under the curve (AUC) bronchodilator response after Visit 3 methacholine challenge. 2.5mg of albuterol was administered at the time of maximal brochoconstriction once the methacholine PC20 was reached. Participants had received Advair for 2 weeks at Visit 3.
Measure: Mean (Standard Deviation); unit: Liters*min
Groups:
- Whites ADRB2:ARG16ARG; Whites ADRB2:GLY16GLY; African Americans ADRB2:ARG16ARG; African Americans ADRB2:GLY16GLY: All participants who had received Advair for 2 weeks at Visit 3.
Arm/Group | Whites ADRB2:ARG16ARG | Whites ADRB2:GLY16GLY | African Americans ADRB2:ARG16ARG | African Americans ADRB2:GLY16GLY
Number analyzed (Participants) | 18 | 23 | 17 | 22
Liters*min | 183.6 (67.02) | 189.2 (61.08) | 160.0 (48.01) | 157.7 (45.28)

6. Secondary Outcome: Bronchodilator Response Following Methacholine Challenge at Visit 4
Description: The area under the curve (AUC) bronchodilator response after Visit 4 methacholine challenge. 2.5mg of albuterol was administered at the time of maximal brochoconstriction once the methacholine PC20 was reached and the change in FEV1 was measured over the next 60 minutes post albuterol administration (bronchodilator response). FEV1 was measured at the following times: 0 (immediately upon completion of nebulization) and at 1, 3, 5, 10, 15, 20, 30, 45, and 60 minutes. Participants had discontinued Advair for 36 hours.
Time Frame: 0 (immediately upon completion of nebulization) and at 1, 3, 5, 10, 15, 20, 30, 45, and 60 minutes after nebulization was complete which occurred 36 hours after the last dose of Advair
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Liters*min
Groups:
- Whites ADRB2:ARG16ARG; Whites ADRB2:GLY16GLY; African Americans ADRB2:ARG16ARG; African Americans ADRB2:GLY16GLY: Participants had discontinued Advair for 36 hours.
Arm/Group | Whites ADRB2:ARG16ARG | Whites ADRB2:GLY16GLY | African Americans ADRB2:ARG16ARG | African Americans ADRB2:GLY16GLY
Number analyzed (Participants) | 18 | 21 | 17 | 22
Liters*min | 187.3 (66.17) | 187.1 (58.31) | 163.2 (46.70) | 157.7 (36.44)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the study period from Visit 1 through Visit 4 (approximately 4 weeks total follow-up).
Arm/Group | Whites ADRB2:ARG16ARG | Whites ADRB2:GLY16GLY | African American ADRB2:ARG16ARG | African American ADRB2:GLY16GLY
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/26 | 0/18 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/26 | 0/18 | 0/25
Other Adverse Events (participants affected / at risk) | 0/19 | 1/26 | 0/18 | 0/25
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Whites ADRB2:ARG16ARG (N=19) | Whites ADRB2:GLY16GLY (N=26) | African American ADRB2:ARG16ARG (N=18) | African American ADRB2:GLY16GLY (N=25)
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant developed worsening asthma after methacholine challenge at Visit 2. The PCP started the participant on prednisone and oxygen.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No